CLINICAL TRIAL: NCT00907153
Title: Vitamin D Supplementation in Polycystic Ovary Syndrome: a Randomized Controlled Trial.
Brief Title: Vitamin D for the Treatment of Women With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Nazia Raja-Khan, M.D., Assistant Professor of Medicine, Division of Endocrinology, Diabetes, and Metabolism, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 29714
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-11

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Vitamin D; Insulin resistance; Inflammation
MeSH Terms: conditions — Polycystic Ovary Syndrome; Insulin Resistance; Inflammation | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental)
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D 300 mcg by mouth once daily for 12 weeks
  Arms: Vitamin D
Drug: Placebo — Placebo by mouth once daily for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if vitamin D will improve insulin resistance, inflammation, and overall well-being in women with PCOS.

DETAILED DESCRIPTION:
As many cells throughout the body possess the vitamin D receptor, adequate vitamin D levels may be essential for multiple physiologic functions. In recent years, vitamin D insufficiency has been linked to insulin resistance, inflammation, poor psychological health, obesity, type 2 diabetes, and cardiovascular disease - these are also commonly found in women with Polycystic Ovary syndrome (PCOS). We believe that vitamin D insufficiency contributes to insulin resistance, inflammation, and psychological distress in women with PCOS. These adverse effects may ultimately increase the risk for serious long-term complications in PCOS, including type 2 diabetes and cardiovascular disease. The key objectives of this research study are to determine the effects of vitamin D supplementation on insulin resistance, inflammation, mood and overall well-being in women with PCOS.

The protocol has been modified by adding the following specific aim: To compare vascular function in healthy age and BMI similar matched women to PCOS women pre-treatment. Our hypothesis is that PCOS women will have greater attenuations in retinal vascular reactivity compared to healthy control women, demonstrating poorer endothelial function. We are currently recruiting healthy women who are age and BMI similar to the PCOS women and measure their retinal vascular reactivity for comparisons to the PCOS women's pre-treatment vascular reactivity. These healthy women will only have a baseline visit in which retinal vascular reactivity will be measured. They will not be enrolled in the placebo or Vitamin D randomization process as described above.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS based on:

  * Eight or fewer menstrual periods per year or spontaneous intermenstrual periods of greater than or equal to 45 days, and
  * Elevated testosterone levels

Exclusion Criteria:

* Current Pregnancy or Nursing
* Elevated calcium
* Kidney Stones or kidney disease
* Current use of vitamin D (other than a multivitamin)
* Use of metformin or other insulin sensitizing drugs in the last 3 months
* Elevated prolactin or untreated thyroid disease
* Diabetes, Liver disease, Heart disease, or other serious medical condition

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-05; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nazia Raja-Khan, M.D., Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Result] Raja-Khan N, Shah J, Stetter CM, Lott ME, Kunselman AR, Dodson WC, Legro RS. High-dose vitamin D supplementation and measures of insulin sensitivity in polycystic ovary syndrome: a randomized, controlled pilot trial. Fertil Steril. 2014 Jun;101(6):1740-6. doi: 10.1016/j.fertnstert.2014.02.021. Epub 2014 Mar 14. PMID 24636395

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 patients were screened for eligibility between July 2009 and November 2010 at Medicine and Obstetrics and Gynecology clinics at an academic medical center in Hershey, PA.
Pre-assignment Details: 28 of 36 participants were randomized. Of those not randomized, 3 did not meet inclusion criteria, 3 declined to participate, and 2 were not randomized for other reasons.
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 13 | 15
Completed | 11 | 11
Not Completed | 2 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (5.2) | 28.7 (5.6) | 28.5 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 14 | 24
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 37.20 (4.53) | 35.09 (9.81) | 36.1 (7.8)
Systolic blood pressure [Mean (Standard Deviation); unit: mm Hg] | 117.46 (10.00) | 113.91 (10.21) | 115.56 (10.11)
Diastolic blood pressure [Mean (Standard Deviation); unit: mm hg] | 79.08 (8.28) | 74.88 (7.72) | 76.83 (7.98)
25-hydroxyvitamin D [Mean (Standard Deviation); unit: ng/mL] | 19.95 (9.47) | 22.20 (6.86) | 21.15 (8.10)
Vitamin D binding protein [Mean (Standard Deviation); unit: mg/dL] | 30.46 (8.53) | 31.95 (7.54) | 31.34 (8.04)
Intact parathyroid hormone (i-PTH) [Mean (Standard Deviation); unit: pg/mL] | 40.81 (27.34) | 33.17 (17.73) | 36.72 (22.19)
Fasting glucose [Mean (Standard Deviation); unit: mg/dL] | 84.92 (9.46) | 83.73 (9.33) | 84.29 (9.23)
Fasting insulin [Mean (Standard Deviation); unit: uU/mL] | 26.31 (9.60) | 27.13 (15.79) | 26.75 (13.05)
2-hour glucose [Mean (Standard Deviation); unit: mg/dL] | 122.08 (36.29) | 110.07 (23.68) | 115.64 (30.22)
2-hour insulin [Mean (Standard Deviation); unit: uU/mL] | 214.69 (146.41) | 107.07 (55.20) | 157.04 (118.72)
Insulin sensitivity index 0,120 [Mean (Standard Deviation); unit: mg·l^2/mmol·mU·min] — Participants underwent a 75-g oral glucose tolerance test, in which blood samples for glucose and insulin were obtained at 0 and 120 minutes and used to calculate the insulin sensitivity index (ISI0,120). The ISI 0,120 = the glucose uptake rate divided by the mean plasma glucose divided by the log(mean serum insulin).
  mg·l^2/mmol·mU·min | 55.55 (23.26) | 63.56 (16.37) | 59.84 (19.57)
Quantitative Insulin Sensitivity Check Index (QUICKI) [Mean (Standard Deviation); unit: units on a scale] — The primary outcome was quantitative insulin sensitivity check index (QUICKI), a validated measure of insulin sensitivity based on fasting insulin and glucose. Quantitative insulin sensitivity check index (QUICKI) = 1/[log(I(0)) + log(G(0))]).
  units on a scale | 0.302 (0.014) | 0.307 (0.029) | 0.305 (0.022)
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) [Mean (Standard Deviation); unit: units on a scale] — HOMA-IR is calculated as the product of fasting glucose and insulin divided by 22.5.
  units on a scale | 5.47 (1.82) | 5.80 (3.90) | 5.65 (2.93)
Total cholesterol [Mean (Standard Deviation); unit: mg/dL] | 172.00 (42.70) | 184.27 (32.52) | 178.57 (37.38)
HDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 45.54 (17.60) | 37.00 (10.83) | 40.96 (14.74)
LDL cholesterol [Mean (Standard Deviation); unit: mg/dL] | 98.62 (36.96) | 117.33 (28.56) | 108.64 (33.47)
Triglyecrides [Mean (Standard Deviation); unit: mg/dL] | 139.08 (71.61) | 149.47 (85.46) | 144.64 (78.07)
High sensitive C-reactive protein (hsCRP) [Mean (Standard Deviation); unit: mg/L] | 7.95 (5.24) | 4.42 (4.34) | 6.1 (5.0)
Total testosterone [Mean (Standard Deviation); unit: ng/dL] | 54.23 (28.16) | 41.27 (17.29) | 48.48 (23.03)
Free testosterone [Mean (Standard Deviation); unit: ng/dL] | 19.08 (15.79) | 14.00 (10.88) | 16.89 (13.33)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Quantitative Insulin Sensitivity Check Index (QUICKI)
Description: Quantitative insulin sensitivity check index (QUICKI) is a validated measure of insulin sensitivity based on fasting insulin and glucose. Quantitative insulin sensitivity check index (QUICKI) = 1/[log(I(0)) + log(G(0))]).
Time Frame: Baseline and 12 weeks
Population: All analyses were by intention to treat. All randomized participants received and ingested the treatment that they were randomly assigned to.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
units on a scale | -0.008 [-0.020 to 0.004] | 0.009 [-0.003 to 0.021]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.05, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = -0.017, 95% CI 2-sided [-0.034 to -0.000]

2. Secondary Outcome: Change From Baseline in Mean High Sensitive C-reactive Protein (hsCRP)
Description: High sensitive C-reactive protein (hsCRP) was assessed as a measure of inflammation.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/L
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mg/L | 0.90 [-2.46 to 4.27] | 2.04 [-1.37 to 5.45]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.62, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = -1.14, 95% CI 2-sided [-5.89 to 3.62]

3. Secondary Outcome: Change From Baseline in Mean Systolic Blood Pressure
Description: Blood pressure was measured in the right arm in the sitting position after a 15-minute rest.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mm Hg | 0.64 [-7.13 to 8.42] | 4.29 [-3.15 to 11.74]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.48, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = -3.65, 95% CI 2-sided [-14.32 to 7.02]

4. Secondary Outcome: Change From Baseline in Mean Diastolic Blood Pressure
Description: Blood pressure was measured in the right arm in the sitting position after a 15-minute rest.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mm Hg | -0.91 [-4.96 to 3.14] | 5.60 [1.69 to 9.52]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.02, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = -6.51, 95% CI 2-sided [-12.07 to -0.96]

5. Secondary Outcome: Change From Baseline in Mean Fasting Glucose
Description: Glucose was assessed after 12 hours of fasting.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mg/dL | -0.70 [-7.96 to 6.56] | -6.98 [-14.31 to 0.34]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.22, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = 6.28, 95% CI 2-sided [-3.97 to 16.54]

6. Secondary Outcome: Change From Baseline in Mean Fasting Insulin
Description: Insulin was assessed after 12 hours of fasting.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: uU/mL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
uU/mL | 13.04 [-3.96 to 30.05] | -0.80 [-18.03 to 16.43]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.33, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = 13.84, 95% CI 2-sided [-210.29 to 37.98]

7. Secondary Outcome: Change From Baseline in Mean 2-hour Glucose
Description: Participants underwent a 75-gram oral glucose tolerance test, in which blood samples for glucose and insulin were obtained at 0 and 2 hours and used to calculate the insulin sensitivity index (ISI 0,120).
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mg/dL | -11.66 [-33.22 to 9.89] | 1.14 [-20.10 to 22.38]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.39, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = -12.80, 95% CI 2-sided [-42.94 to 17.34]

8. Secondary Outcome: Change From Baseline in Mean 2-hour Insulin
Description: as for outcome 7
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: uU/mL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
uU/mL | -62.02 [-124.5 to 0.49] | 13.06 [-47.94 to 74.06]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.09, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = -75.08, 95% CI 2-sided [-161.9 to 11.78]

9. Secondary Outcome: Change From Baseline in Mean Insulin Sensitivity Index (ISI 0,120)
Description: Participants underwent a 75-g oral glucose tolerance test, in which blood samples for glucose and insulin were obtained at 0 and 120 minutes and used to calculate the insulin sensitivity index (ISI0,120). The ISI 0,120 = the glucose uptake rate divided by the mean plasma glucose divided by the log(mean serum insulin).
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg·l^2/mmol·mU·min
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mg·l^2/mmol·mU·min | 6.67 [-16.87 to 30.21] | 5.94 [-17.77 to 29.65]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.96, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = 0.73, 95% CI 2-sided [-32.59 to 34.06]

10. Secondary Outcome: Change From Baseline in Mean Homeostatic Model Assessment of Insulin Resistance (HOMA-IR)
Description: Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) is a validated measure of insulin resistance based on fasting insulin and glucose. HOMA-IR is calculated as the product of fasting glucose and insulin divided by 22.5.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
units on a scale | 2.57 [-0.90 to 6.03] | -0.51 [-4.01 to 2.99]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.21, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = 3.08, 95% CI 2-sided [-1.84 to 7.99]

11. Secondary Outcome: Change From Baseline in Mean Total Cholesterol
Description: Lipid profile was assessed after 12 hours of fasting.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mg/dL | -1.69 [-19.04 to 15.66] | -1.80 [-19.55 to 15.95]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.99, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = 0.11, 95% CI 2-sided [-24.43 to 24.64]

12. Secondary Outcome: Change From Baseline in Mean HDL Cholesterol
Description: Lipid profile was assessed after 12 hours of fasting.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mg/dL | -0.70 [-6.52 to 5.12] | 1.23 [-4.68 to 7.14]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.62, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Median Difference (Net) = -1.93, 95% CI 2-sided [-10.12 to 6.26]

13. Secondary Outcome: Change From Baseline in Mean LDL Cholesterol
Description: Lipid profile was assessed after 12 hours of fasting.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mg/dL | -0.12 [-14.70 to 14.46] | -0.40 [-15.24 to 14.45]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.98, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = 0.28, 95% CI 2-sided [-20.29 to 20.85]

14. Secondary Outcome: Change From Baseline in Mean Triglycerides
Description: Lipid profile was assessed after 12 hours of fasting.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mg/dL | -2.21 [-34.11 to 29.69] | -12.44 [-44.68 to 19.80]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.64, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = 10.24, 95% CI 2-sided [-34.61 to 55.08]

15. Secondary Outcome: Change From Baseline in Mean Total Testosterone
Description: Total and free testosterone levels were assessed from blood samples to evaluate effects on hyperandrogenemia in PCOS.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ng/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
ng/dL | 3.01 [-8.05 to 14.06] | 10.16 [-1.16 to 21.47]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.88, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = 0.88, 95% CI 2-sided [-22.81 to 8.51]

16. Secondary Outcome: Change From Baseline in Mean Free Testosterone
Description: Total and free testosterone levels were assessed from blood samples to evaluate effects on hyperandrogenemia in PCOS.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ng/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
ng/dL | 2.67 [-1.29 to 6.63] | 5.82 [1.82 to 9.82]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.25, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = -3.15, 95% CI 2-sided [-8.70 to 2.41]

17. Other Pre Specified Outcome: Change From Baseline in Mean 25-hydroxyvitamin D
Description: Total 25-hydroxyvitamin D was assayed by the Immunodiagnostic Systems radioimmunoassay.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
ng/mL | 45.63 [33.50 to 57.76] | 1.32 [-10.93 to 13.58]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p < 0.001, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = 44.31, 95% CI 2-sided [27.13 to 61.48]

18. Other Pre Specified Outcome: Change From Baseline in Mean Vitamin D Binding Protein
Description: Vitamin D binding protein levels were assessed as it has been linked with insulin resistance and type 2 diabetes.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
mg/dL | 1.01 [-1.60 to 3.62] | -0.55 [-3.14 to 2.04]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.38, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = 1.56, 95% CI 2-sided [-2.08 to 5.20]

19. Other Pre Specified Outcome: Change From Baseline in Mean Intact Parathyroid Hormone (i-PTH)
Description: Intact parathyroid hormone levels were assessed as they have been linked with obesity and insulin resistance.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: pg/mL
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 13 | 15
pg/mL | -24.28 [-39.80 to -8.76] | -16.45 [-31.40 to -1.49]
Statistical Analysis 1: Comparison: Vitamin D vs Placebo; Test type: Superiority; p = 0.46, Regression, Linear; Model-based differences adjusted for oral contraceptive use and season; Mean Difference (Net) = -7.84, 95% CI 2-sided [-29.34 to 13.67]

ADVERSE EVENTS:
Time Frame: Twelve weeks.
Arm/Group | Vitamin D | Placebo
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes